CLINICAL TRIAL: NCT03734822
Title: Comparative Analysis of CO2 Monitoring Methods in Patients With CF Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Anne May, Assistant Professor of Clinical Pediatrics, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB15-00797
Record Dates: First submitted 2018-10-23; First posted 2018-11-08 (Actual); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CF (Other): Cystic fibrosis patients undergoing general anesthesia.
  Interventions: Other: End tidal CO2 (EtCO2); Device: Transcutaneous CO2 (TCO2); Diagnostic Test: Capillary CO2 (CapCO2); Diagnostic Test: Arterial blood gas (ABG)

INTERVENTIONS:
Other: End tidal CO2 (EtCO2) — End tidal CO2 (EtCO2) is monitored through the endotracheal tube during general anesthesia.
Device: Transcutaneous CO2 (TCO2) — Continuous and noninvasive real-time monitoring of transcutaneous CO2.
  Other Names: The SenTec Digital Monitoring System (SDMS)
Diagnostic Test: Capillary CO2 (CapCO2) — Capillary CO2 collected by finger stick and run on the i-STAT handheld blood analyzer.
Diagnostic Test: Arterial blood gas (ABG) — Arterial blood gas collected from the radial artery and run on the i-STAT handheld blood analyzer.

SUMMARY:
Four methods are routinely used to monitor CO2 in patients. End tidal CO2 (EtCO2) is monitored through the endotracheal tube during general anesthesia. CO2 is also monitored in other healthcare settings transcutaneously (TCO2), via finger stick capillary CO2 (CapCO2), and arterial blood gas (ABG). The purpose of this study is to perform all four measurements simultaneously during general anesthesia to identify which measure provides the most accurate data with the least amount of patient risk.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of cystic fibrosis (positive sweat chloride value ≥ 60 mEq/L) and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with the CF phenotype)
* Hemodynamically stable undergoing general anesthesia for a scheduled procedure

Exclusion Criteria:

* Patients not diagnosed with CF
* CF patients undergoing anesthesia for emergency procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystic Fibrosis: Cystic fibrosis patients undergoing general anesthesia.
  End tidal CO2 (EtCO2): End tidal CO2 (EtCO2) is monitored through the endotracheal tube during general anesthesia.
  Transcutaneous CO2 (TCO2): Continuous and noninvasive real-time monitoring of transcutaneous CO2.
  Capillary CO2 (CapCO2): Capillary CO2 collected by finger stick and run on the i-STAT handheld blood analyzer.
  Arterial blood gas (ABG): Arterial blood gas collected from the radial artery and run on the i-STAT handheld blood analyzer.
Period: Overall Study
Arm/Group | Cystic Fibrosis
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cystic Fibrosis
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 47
BMI (kg/m2) [Median (Inter-Quartile Range); unit: Kg/m2] | 18.7 [16.7 to 21.4]
FEV1% [Mean (Standard Deviation); unit: percentage of normal] — FEV1 is the maximal amount of air you can forcefully exhale in one second. It is then converted to a percentage of normal.
  FEV1 greater 80% of predicted= normal, FEV1 60% to 79% of predicted = Mild obstruction, FEV1 40% to 59% of predicted = Moderate obstruction, FEV1 less than 40% of predicted = Severe obstruction
  percentage of normal | 87.3 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CO2 Levels
Description: Looking at the accuracy of CO2 levels assessed via end tidal CO2 (ETCO2), capillary CO2 (Cap-CO2), and transcutaneous CO2 (TCCO2) compared to arterial blood gas (ABG) which is the gold standard.
Time Frame: Immediately following induction of anesthesia
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cystic Fibrosis
Number analyzed (Participants) | 47
mmHg
  PaCO2 from ABG | 48.9 (7.9)
  ETCO2 | 39.5 (6.2)
  TCCO2 | 41.5 (9.4)
  Cap-CO2 | 44.3 (8.6)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Cystic Fibrosis
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03734822/Prot_SAP_000.pdf